CLINICAL TRIAL: NCT01869712
Title: Using Partially Randomized Patient Preference Research Model for Evaluation the Therapeutic Effect of Non-pharmaceutical Therapies: Protocol for a Feasibility Study
Brief Title: PRPP Model for Evaluation the Effect of Non-pharmaceutical Therapies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huijuan Cao, Research Associate, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0100604024
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Fibromyalgia
Keywords: cupping therapy; acupuncture; partially randomized; patient preference; fibromyalgia; criteria formulated by American College Rheumatology 2002
MeSH Terms: conditions — Fibromyalgia; Patient Preference | interventions — Cupping Therapy; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cupping therapy (randomized) (Experimental): Use retained cupping as the main cupping method, supplemented with flash cupping and/or moving cupping. First use empty cupping, which means the cups are removed after suction without delay, then practitioners should control the suction by gently moving the cup toward direction of DU and/or BL, repeat this moving for several times, finally cupping practitioners utilize the flaming heating power to achieve suction (minus pressure) inside the cups to make them apply on the desired part of the body. Cups should retain for 10 minutes daily, patients accept the treatment three times weekly for totally 15 times.
  Interventions: Other: Cupping therapy
- Cupping therapy (non-randomized) (Experimental): Use retained cupping as the main cupping method, supplemented with flash cupping and/or moving cupping. First use empty cupping, which means the cups are removed after suction without delay, then practitioners should control the suction by gently moving the cup toward direction of DU and/or BL, repeat this moving for several times, finally cupping practitioners utilize the flaming heating power to achieve suction (minus pressure) inside the cups to make them apply on the desired part of the body. Cups should retain for 10 minutes daily, patients accept the treatment three times weekly for totally 15 times.
  Interventions: Other: Cupping therapy
- Acupuncture (non-randomized) (Active Comparator): Sterilize the selected points with alcohol, and then select the specific size of needles to do the acupuncture. Do the manual stimulation for seconds after needles' insertion, including twist, pull up and deeper insert. Needles should be withdrawn after 30 minutes. Patients accept the treatment three times weekly for totally 15 times.
  Interventions: Other: Acupuncture
- Acupuncture (randomized) (Active Comparator): Sterilize the selected points with alcohol, and then select the specific size of needles to do the acupuncture. Do the manual stimulation for seconds after needles' insertion, including twist, pull up and deeper insert. Needles should be withdrawn after 30 minutes.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Cupping therapy
  Arms: Cupping therapy (non-randomized); Cupping therapy (randomized)
Other: Acupuncture
  Arms: Acupuncture (non-randomized); Acupuncture (randomized)

SUMMARY:
To assess the application of partially randomized patient preference (PRPP) trial model which concerns the patients' preference on evaluation the therapeutic effect of non-pharmaceutical therapy, and to observe the therapeutic effect of two kinds of non-pharmaceutical therapies (acupuncture and cupping therapy) for fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fibromyalgia diagnosed according to criteria formulated by American College Rheumatology 2002;
* Patients whose scores for pain intensity is more than 30mm;
* Patients who are 20 to 60 years old;
* Patients who fully understand the process of this research and who are willing to provide informed consent.

Exclusion Criteria:

* The widespread muscular-skeletal pain is caused by some kind of disease, surgery, or other external interference factors (except fibromyalgia);
* Patients with mental disorders, or other serious organic diseases, such as organ failure;
* Patients who take oral anodyne medications or accept other interventions for pain relief during the treatment;
* Pregnant or lactating women;
* Patients currently participating in another clinical trial.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Patients' compliance | Record the number of drop out or lost during the 5 weeks' treatment and 3 months' follow up duration (for an expected totally 17 weeks) and note the reason for missing data
Patients satisfactory for the treatment | The satisfactory for the treatment is investigated at week 5 (as the end of the treatment).
  Satisfactory for the treatment is measured by a seven-score scale, with 1 for "very satisfied" and 7 for "very unsatisfied".
Practitioners' attitude for the research model | Practitioners' attitude for the research model is investigated at week 5 (as the end of the treatment).
  Individual interview or the focus group interview will be applied after the treatment, all the practitioners in the study (including acupuncturists and cupping therapy practitioners) will be interviewed to know their attitude for conducting the partially randomized patient preference trial model and their thoughts of this model compare to general randomized controlled trial.

SECONDARY OUTCOMES:
Adverse events | Adverse events will be observed for the duration of 5 weeks' treatment and 3 months' follow-up, with an expected average of totally 17 weeks.
  Researchers should note any minor or serious adverse event occurs during treatment and follow up duration, including cases and symptoms of patients with adverse events.
Patients' expectation for the treatment | Patients' expectation is investigated at week 0
  Patients' expectation is measured by a four-score scale, with 1 for "symptoms are totally disappear" and 4 for "no change for symptoms".
Visual Analogue Scale (VAS) for pain intensity | VAS should be measured seven times at week 0, the end of each five times treatment (totally fifteen times treatment in 5 weeks), week 9, week 13, and week 17, respectively.
  The length of scale of VAS is 100mm, 0 is representing for no pain, and 100 is representing unbearable pain which may affect appetite and quality of sleep. Researchers should show the scale to patients, and note the scores of pain degree given by patients according to the scale.

OTHER OUTCOMES:
Widespread Pain Index (WPI）for pain intensity | WPI should be measured seven times at week 0, the end of each five times treatment (totally fifteen times treatment in 5 weeks), week 9, week 13, and week 17, respectively.
  WPI is defined according to the American College of Rheumatology diagnostic criteria （2002）for fibromyalgia.
Symptom Severity (SS) for pain intensity | SS should be measured seven times at week 0, the end of each five times treatment (totally fifteen times treatment in 5 weeks), week 9, week 13, and week 17, respectively.
  SS is defined according to the American College of Rheumatology diagnostic criteria （2002）for fibromyalgia
Hamilton Depression Scale (HAMD) | HAMD is measured totally 3 times at week 0, week 5 and week 17, respectively.
Quality of life measured by The Medical Outcome Study 36-item short-form health survey (SF36) | SF36 is measured totally 3 times at week 0, week 5 and week 17, respectively.
Fibromyalgia Intensive Questionnaire (FIQ) | FIQ is measured totally 3 times at week 0, week 5 and week 17, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Huijuan Cao, Ph.D., Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- Beijing University of Chinese Medicine Affiliated Dongfang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Cao H, Hu H, Colagiuri B, Liu J. Medicinal cupping therapy in 30 patients with fibromyalgia: a case series observation. Forsch Komplementmed. 2011;18(3):122-6. doi: 10.1159/000329329. Epub 2011 May 24. PMID 21701180
- [Background] Cao H, Liu J, Lewith GT. Traditional Chinese Medicine for treatment of fibromyalgia: a systematic review of randomized controlled trials. J Altern Complement Med. 2010 Apr;16(4):397-409. doi: 10.1089/acm.2009.0599. PMID 20423209
- [Derived] Cao HJ, Liu JP, Hu H, Wang NS. Using a partially randomized patient preference study design to evaluate the therapeutic effect of acupuncture and cupping therapy for fibromyalgia: study protocol for a partially randomized controlled trial. Trials. 2014 Jul 10;15:280. doi: 10.1186/1745-6215-15-280. PMID 25012121